CLINICAL TRIAL: NCT00655876
Title: A Phase III Trial Evaluating the Addition of Cetuximab to Paclitaxel, Cisplatin, and Radiation for Patients With Esophageal Cancer Who Are Treated Without Surgery
Brief Title: Paclitaxel, Cisplatin, and Radiation Therapy With or Without Cetuximab in Treating Patients With Locally Advanced Esophageal Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RTOG 0436; CDR0000538085
Record Dates: First submitted 2008-04-09; First posted 2008-04-10 (Estimated); Results first posted 2018-03-14 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-05

CONDITIONS: Esophageal Cancer
Keywords: stage IIA esophageal cancer; stage IIB esophageal cancer; stage IIIA esophageal cancer; stage IIIB esophageal cancer; stage IIIC esophageal cancer; stage IV esophageal cancer; squamous cell carcinoma of the esophagus
MeSH Terms: conditions — Esophageal Neoplasms; Esophageal Squamous Cell Carcinoma | interventions — Cetuximab; Cisplatin; Paclitaxel; Radiotherapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Chemoradiation + Cetuximab (Experimental): External beam radiation therapy (RT) with concurrent weekly paclitaxel, cisplatin, and cetuximab
  Interventions: Drug: cetuximab; Drug: cisplatin; Drug: paclitaxel; Radiation: radiation therapy
- Chemoradiation (Active Comparator): External beam radiation therapy with concurrent weekly paclitaxel, and cisplatin
  Interventions: Drug: cisplatin; Drug: paclitaxel; Radiation: radiation therapy

INTERVENTIONS:
Drug: cetuximab — Weekly with external beam radiation therapy for a total of six doses. The initial dose of cetuximab is 400 mg/m^2 intravenously administered over 120 minutes on day 1, followed by weekly infusions of 250 mg/m^2 intravenously over 60 minutes on days 8, 15, 22, 29, and 36. The infusion rate of cetuximab must never exceed 5 mL/min.
  Arms: Chemoradiation + Cetuximab
Drug: cisplatin — Weekly with external beam radiation therapy for a total of six doses. Patients receive 25 mg/m^2 as an intravenous infusion over 30-60 minutes on days 1, 8, 15, 22, 29 and 36.
Drug: paclitaxel — Weekly with external beam radiation therapy for a total of six doses. Patients receive 50 mg/m^2 as an intravenous infusion over 1 hour on days 1, 8, 15, 22, 29 and 36.
Radiation: radiation therapy — 1.8 Gy daily for 28 days (over 5-6 weeks) for a total dose of 50.4 Gy.

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as paclitaxel and cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to kill tumor cells. Monoclonal antibodies, such as cetuximab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Cetuximab may stop the growth of esophageal cancer by blocking blood flow to the tumor. It is not yet known whether giving paclitaxel and cisplatin together with radiation therapy is more effective with or without cetuximab in treating esophageal cancer.

PURPOSE: This randomized phase III trial is comparing how well giving paclitaxel and cisplatin together with radiation therapy works with or without cetuximab in treating patients with locally advanced esophageal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate whether the addition of cetuximab to chemotherapy comprising paclitaxel, cisplatin, and radiotherapy improves overall survival compared with paclitaxel, cisplatin, and radiotherapy alone in patients with esophageal cancer treated without surgery.

Secondary

* To evaluate whether the addition of cetuximab to paclitaxel, cisplatin, and radiotherapy improves local control by increasing the clinical complete response and decreasing local recurrence in these patients.
* To evaluate adverse events in these patients.
* To evaluate endoscopic complete response rates in these patients.
* To evaluate if the addition of cetuximab to paclitaxel, cisplatin, and radiotherapy improves the Esophageal Cancer Subscale (ECS) score of the Functional Assessment of Cancer Therapy - Esophagus (FACT-E) quality of life tool.
* To evaluate the quality-adjusted survival of each treatment arm using EQ-5D if the primary endpoint supports the primary hypothesis.

OUTLINE: This is a multicenter study. Patients are stratified according to histology (adenocarcinoma vs squamous), cancer lesion size (< 5 cm vs ≥ 5 cm), and disease status of celiac nodes (present vs absent). Patients are randomized to 1 of 2 treatment arms.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically (histologic or cytologic) proven diagnosis of primary squamous cell or adenocarcinoma of the esophagus or gastroesophageal junction within 12 weeks prior to registration. Patients with involvement of the gastroesophageal junction with Siewert type I or II tumors (tumors arising from the distal esophagus and involving the esophagogastric junction or tumors starting at the esophagogastric junction and involving the cardia) are eligible.

   * 1.1 Disease must be encompassed in a radiotherapy field.
   * 1.2 Patients with celiac, perigastric, mediastinal or supraclavicular adenopathy are eligible.
   * 1.3 Patients with cervical esophageal carcinoma are eligible.
2. Stage T1N1M0; T2-4, Any N, M0; Any T, Any N, M1a, based upon the following minimum diagnostic work-up:

   * 2.1 History/physical examination within 6 weeks prior to registration
   * 2.2 Positron emission tomography (PET)/positron emission tomography-computed tomography (PET-CT) scan (strongly recommended) or chest/abdominal CT within 6 weeks prior to registration
   * 2.3 Electrocardiogram (EKG) within 6 weeks of study entry
   * 2.4 Endoscopy with biopsy or cytology by fine needle aspiration (FNA) (must be able to document histologic subtype) within 12 weeks of study entry. Patients with T3-4 proximal thoracic esophageal tumors (15-25 cm) must undergo bronchoscopy to exclude fistula. (NOTE: Any images from endoscopic procedures up to the time of progression must be kept in the patient's confidential study file.)
3. Zubrod performance status 0-2
4. Age ≥ 18 and ≤ 74 (upper limit was set at 74 in an amendment)
5. Complete blood count (CBC)/differential obtained within 2 weeks prior to registration on study, with adequate bone marrow function defined as follows:

   * 5.1 Absolute neutrophil count (ANC) ≥ 1,500 cells/mm3
   * 5.2 Platelets ≥ 100,000 cells/mm3
   * 5.3 Hemoglobin ≥ 8.0 g/dl (Note: The use of transfusion or other intervention to achieve Hgb ≥8.0 g/dl is acceptable.)
6. Additional laboratory studies obtained within 2 weeks prior to registration on study

   * 6.1 Creatinine ≤ 1.5 mg/dl
   * 6.2 Bilirubin ≤ 1.5 x upper limit of normal
   * 6.3 Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) ≤ 3 x upper limit of normal
   * 6.4 Serum pregnancy test for women of childbearing potential
7. Patient's total intake (oral/enteral) must be ≥ 1500 kCal/day
8. Patient must provide study-specific informed consent prior to study entry
9. Women of childbearing potential and male participants must practice adequate contraception

Exclusion Criteria:

1. Evidence of tracheoesophageal fistula, or invasion into the trachea or major bronchi. Patients with T3-4 proximal thoracic esophageal tumors (15-25 cm) must undergo bronchoscopy to exclude fistula.
2. Prior invasive malignancy (except non-melanomatous skin cancer) unless disease free for a minimum of 2 years (For example, carcinoma in situ of the breast, oral cavity, or cervix are all permissible).
3. Prior systemic chemotherapy for esophageal cancer; note that prior chemotherapy for a different cancer is allowable.
4. Prior radiation therapy that would result in overlap of planned radiation therapy fields.
5. Prior therapy that specifically and directly targets the epidermal growth factor receptor (EGFR) pathway.
6. Prior platinum-based and/or paclitaxel-based therapy.
7. Prior allergic reaction to the study drugs involved in this protocol.
8. Prior severe infusion reaction to a monoclonal antibody.
9. Severe, active comorbidity, defined as follows:

   * 9.1 Unstable angina and/or congestive heart failure requiring hospitalization within the last 3 months
   * 9.2 Transmural myocardial infarction within the last 6 months
   * 9.3 Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration
   * 9.4 Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy at the time of registration
   * 9.5 Acquired immune deficiency syndrome (AIDS) based upon current Centers for Disease Control and Prevention (CDC) definition; note, however, that human immunodeficiency virus (HIV) testing is not required for entry into this protocol. The need to exclude patients with AIDS from this protocol is necessary because the treatments involved in this protocol may be significantly immunosuppressive. Protocol-specific requirements may also exclude immunocompromised patients.
10. Pregnancy or women of childbearing potential and men who are sexually active and not willing/able to use medically acceptable forms of contraception; this exclusion is necessary because the treatment involved in this study may be significantly teratogenic.
11. Women who are nursing.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 344 (Actual)
Dates: Start 2008-06; Primary Completion 2015-04 (Actual); Study Completion 2022-05-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mohan Suntharalingam, MD, Principal Investigator — University of Maryland Greenebaum Cancer Center; David H. Ilson, MD, PhD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (175):
- United States (173):
  - Arizona Oncology - Tucson, Tucson, Arizona
  - Auburn Radiation Oncology, Auburn, California
  - Radiation Oncology Centers - Cameron Park, Cameron Park, California
  - Mercy Cancer Center at Mercy San Juan Medical Center, Carmichael, California
  - Enloe Cancer Center at Enloe Medical Center, Chico, California
  - California Cancer Center - Woodward Park Office, Fresno, California
  - Saint Agnes Cancer Center at Saint Agnes Medical Center, Fresno, California
  - Memorial Medical Center, Modesto, California
  - Radiation Oncology Center - Roseville, Roseville, California
  - Radiological Associates of Sacramento Medical Group, Incorporated, Sacramento, California
  - University of California Davis Cancer Center, Sacramento, California
  - Mercy General Hospital, Sacramento, California
  - Solano Radiation Oncology Center, Vacaville, California
  - Sutter Solano Medical Center, Vallejo, California
  - Rocky Mountain Cancer Centers - Aurora, Aurora, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - George Bray Cancer Center at the Hospital of Central Connecticut - New Britain Campus, New Britain, Connecticut
  - William W. Backus Hospital, Norwich, Connecticut
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - University of Florida Shands Cancer Center, Gainesville, Florida
  - Ella Milbank Foshay Cancer Center at Jupiter Medical Center, Jupiter, Florida
  - Center for Cancer Care and Research at Watson Clinic, LLP, Lakeland, Florida
  - Baptist-South Miami Regional Cancer Program, Miami, Florida
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - M.D. Anderson Cancer Center at Orlando, Orlando, Florida
  - John B. Amos Cancer Center, Columbus, Georgia
  - Nancy N. and J. C. Lewis Cancer and Research Pavilion at St. Joseph's/Candler, Savannah, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - Queen's Cancer Institute at Queen's Medical Center, Honolulu, Hawaii
  - Hawaii Medical Center - East, Honolulu, Hawaii
  - Saint Alphonsus Cancer Care Center at Saint Alphonsus Regional Medical Center, Boise, Idaho
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Cardinal Bernardin Cancer Center at Loyola University Medical Center, Maywood, Illinois
  - Advocate Lutheran General Cancer Care Center, Park Ridge, Illinois
  - Swedish-American Regional Cancer Center, Rockford, Illinois
  - Cancer Institute at St. John's Hospital, Springfield, Illinois
  - Saint John's Cancer Center at Saint John's Medical Center, Anderson, Indiana
  - Bloomington Hospital Regional Cancer Institute, Bloomington, Indiana
  - Radiation Oncology Associates Southwest, Fort Wayne, Indiana
  - Parkview Regional Cancer Center at Parkview Health, Fort Wayne, Indiana
  - Methodist Cancer Center at Methodist Hospital, Indianapolis, Indiana
  - Central Indiana Cancer Centers - East, Indianapolis, Indiana
  - Cancer Center at Ball Memorial Hospital, Muncie, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - McFarland Clinic, PC, Ames, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - North Iowa, Mason City, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - Mary Bird Perkins Cancer Center - Baton Rouge, Baton Rouge, Louisiana
  - Greenebaum Cancer Center at University of Maryland Medical Center, Baltimore, Maryland
  - Greater Baltimore Medical Center Cancer Center, Baltimore, Maryland
  - St. Agnes Hospital Cancer Center, Baltimore, Maryland
  - Hudner Oncology Center at Saint Anne's Hospital - Fall River, Fall River, Massachusetts
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - Josephine Ford Cancer Center at Henry Ford Hospital, Detroit, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Lacks Cancer Center at Saint Mary's Health Care, Grand Rapids, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - St. Mary Mercy Hospital, Livonia, Michigan
  - Mercy Regional Cancer Center at Mercy Hospital, Port Huron, Michigan
  - Seton Cancer Institute at Saint Mary's - Saginaw, Saginaw, Michigan
  - MeritCare Bemidji, Bemidji, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Minnesota Oncology - Maplewood, Maplewood, Minnesota
  - Regions Hospital Cancer Care Center, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - University of Mississippi Cancer Clinic, Jackson, Mississippi
  - Cancer Institute of Cape Girardeau, LLC, Cape Girardeau, Missouri
  - Saint Louis University Cancer Center, St Louis, Missouri
  - Missouri Baptist Cancer Center, St Louis, Missouri
  - David C. Pratt Cancer Center at St. John's Mercy, St Louis, Missouri
  - Billings Clinic - Downtown, Billings, Montana
  - Sletten Cancer Institute at Benefis Healthcare, Great Falls, Montana
  - Methodist Estabrook Cancer Center, Omaha, Nebraska
  - Lakeside Hospital, Omaha, Nebraska
  - CCOP - Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Payson Center for Cancer Care at Concord Hospital, Concord, New Hampshire
  - Seacoast Cancer Center at Wentworth - Douglass Hospital, Dover, New Hampshire
  - Center for Cancer Care at Exeter Hospital, Exeter, New Hampshire
  - Kingsbury Center for Cancer Care at Cheshire Medical Center, Keene, New Hampshire
  - Norris Cotton Cancer Center at Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Elliot Regional Cancer Center at Elliot Hospital, Manchester, New Hampshire
  - Monmouth Medical Center, Long Branch, New Jersey
  - Fox Chase Virtua Health Cancer Program at Virtua Memorial Hospital Marlton, Marlton, New Jersey
  - Frederick R. and Betty M. Smith Cancer Treatment Center, Sparta, New Jersey
  - J. Phillip Citta Regional Cancer Center at Community Medical Center, Toms River, New Jersey
  - Cancer Institute of New Jersey at Cooper - Voorhees, Voorhees Township, New Jersey
  - New York Oncology Hematology, PC at Albany Regional Cancer Care, Albany, New York
  - Lourdes Regional Cancer Center, Binghamton, New York
  - Charles R. Wood Cancer Center at Glens Falls Hospital, Glens Falls, New York
  - Beth Israel Medical Center - Petrie Division, New York, New York
  - St. Luke's - Roosevelt Hospital Center - St.Luke's Division, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center at Phelps Memorial Hospital Center, Sleepy Hollow, New York
  - Mission Hospitals - Memorial Campus, Asheville, North Carolina
  - Alamance Cancer Center at Alamance Regional Medical Center, Burlington, North Carolina
  - Presbyterian Cancer Center at Presbyterian Hospital, Charlotte, North Carolina
  - Kinston Medical Specialists, Kinston, North Carolina
  - CCOP - MeritCare Hospital, Fargo, North Dakota
  - McDowell Cancer Center at Akron General Medical Center, Akron, Ohio
  - Summa Center for Cancer Care at Akron City Hospital, Akron, Ohio
  - Barberton Citizens Hospital, Barberton, Ohio
  - Mercy Cancer Center at Mercy Medical Center, Canton, Ohio
  - Aultman Cancer Center at Aultman Hospital, Canton, Ohio
  - Case Comprehensive Cancer Center, Cleveland, Ohio
  - MetroHealth Cancer Care Center at MetroHealth Medical Center, Cleveland, Ohio
  - Lake/University Ireland Cancer Center, Mentor, Ohio
  - Southwest General Health Center, Middleburg Heights, Ohio
  - UHHS Chagrin Highlands Medical Center, Orange, Ohio
  - Robinson Radiation Oncology, Ravenna, Ohio
  - UHHS Westlake Medical Center, Westlake, Ohio
  - Oklahoma University Cancer Institute, Oklahoma City, Oklahoma
  - Natalie Warren Bryant Cancer Center at St. Francis Hospital, Tulsa, Oklahoma
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Willamette Valley Cancer Center - Eugene, Eugene, Oregon
  - Providence Cancer Center at Providence Portland Medical Center, Portland, Oregon
  - Providence St. Vincent Medical Center, Portland, Oregon
  - UPMC Cancer Center at Beaver Medical Center, Beaver, Pennsylvania
  - UPMC Cancer Center at Jefferson Regional Medical Center, Clairton, Pennsylvania
  - Delaware County Regional Cancer Center at Delaware County Memorial Hospital, Drexel Hill, Pennsylvania
  - Regional Cancer Center - Erie, Erie, Pennsylvania
  - Adams Cancer Center, Gettysburg, Pennsylvania
  - UPMC Cancer Center - Arnold Palmer Pavilion, Greensburg, Pennsylvania
  - Frankford Hospital Cancer Center - Torresdale Campus, Philadelphia, Pennsylvania
  - Albert Einstein Cancer Center, Philadelphia, Pennsylvania
  - UPMC - Shadyside, Pittsburgh, Pennsylvania
  - UPMC Cancer Center at UPMC St. Margaret, Pittsburgh, Pennsylvania
  - UPMC Cancer Center at UPMC Passavant, Pittsburgh, Pennsylvania
  - McGlinn Family Regional Cancer Center at Reading Hospital and Medical Center, Reading, Pennsylvania
  - UPMC Cancer Center at UPMC Northwest, Seneca, Pennsylvania
  - York Cancer Center at Apple Hill Medical Center, York, Pennsylvania
  - Rhode Island Hospital Comprehensive Cancer Center, Providence, Rhode Island
  - Northmain Radiation Oncology, Providence, Rhode Island
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - Cancer Centers of the Carolinas - Faris Road, Greenville, South Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - Cancer Centers of the Carolinas - Seneca, Seneca, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Cancer Centers of the Carolinas - Spartanburg, Spartanburg, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Sanford Cancer Center at Sanford USD Medical Center, Sioux Falls, South Dakota
  - Thompson Cancer Survival Center, Knoxville, Tennessee
  - Harrington Cancer Center, Amarillo, Texas
  - Texas Oncology, PA at Harris Center HEB, Bedford, Texas
  - Texas Oncology, PA at Texas Cancer Center - Denton South, Denton, Texas
  - Klabzuba Cancer Center at Harris Methodist Fort Worth Hospital, Fort Worth, Texas
  - Memorial Hermann Hospital - Memorial City, Houston, Texas
  - Longview Cancer Center, Longview, Texas
  - Joe Arrington Cancer Research and Treatment Center, Lubbock, Texas
  - Cancer Care Centers of South Texas - Northeast, San Antonio, Texas
  - Texas Oncology, PA at Texas Cancer Center - Sherman, Sherman, Texas
  - Texas Oncology, PA at Texas Oncology Cancer Center Sugar Land, Sugar Land, Texas
  - Tyler Cancer Center, Tyler, Texas
  - Texas Oncology, PA - Wichita Falls, Wichita Falls, Texas
  - Jon and Karen Huntsman Cancer Center at Intermountain Medical Center, Murray, Utah
  - Utah Cancer Specialists at UCS Cancer Center, Salt Lake City, Utah
  - Huntsman Cancer Institute at University of Utah, Salt Lake City, Utah
  - Dixie Regional Medical Center - East Campus, St. George, Utah
  - Northwest Cancer Specialists at Vancouver Cancer Center, Vancouver, Washington
  - Schiffler Cancer Center at Wheeling Hospital, Wheeling, West Virginia
  - St. Mary's Hospital Medical Center - Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Bay Area Cancer Care Center at Bay Area Medical Center, Marinette, Wisconsin
  - Veterans Affairs Medical Center - Milwaukee, Milwaukee, Wisconsin
  - Regional Cancer Center at Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Door County Cancer Center at Door County Memorial Hospital, Sturgeon Bay, Wisconsin
  - Waukesha Memorial Hospital Regional Cancer Center, Waukesha, Wisconsin
  - University of Wisconcin Cancer Center at Aspirus Wausau Hospital, Wausau, Wisconsin
- Canada (2):
  - Saint John Regional Hospital, Saint John, New Brunswick
  - McGill Cancer Centre at McGill University, Montreal, Quebec

REFERENCES:
- [Result] Suntharalingam M, Winter K, Ilson D, Dicker AP, Kachnic L, Konski A, Chakravarthy AB, Anker CJ, Thakrar H, Horiba N, Dubey A, Greenberger JS, Raben A, Giguere J, Roof K, Videtic G, Pollock J, Safran H, Crane CH. Effect of the Addition of Cetuximab to Paclitaxel, Cisplatin, and Radiation Therapy for Patients With Esophageal Cancer: The NRG Oncology RTOG 0436 Phase 3 Randomized Clinical Trial. JAMA Oncol. 2017 Nov 1;3(11):1520-1528. doi: 10.1001/jamaoncol.2017.1598. PMID 28687830
- Available data/document: Individual Participant Data Set: NCT00655876 — http://nctn-data-archive.nci.nih.gov/ — Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Chemoradiation + Cetuximab | Chemoradiation
Started | 168 | 176
Completed | 159 (Subjects with data available for the primary analysis are considered to have completed the study.) | 169 (Subjects with data available for the primary analysis are considered to have completed the study.)
Not Completed | 9 | 7
Not completed — Protocol Violation | 9 | 7

BASELINE CHARACTERISTICS:
Population: Eligible patients
Groups:
- Total: Total of all reporting groups
Arm/Group | Chemoradiation + Cetuximab | Chemoradiation | Total
Number analyzed (Participants) | 159 | 169 | 328
Age, Continuous [Median (Full Range); unit: years] | 65 [39 to 87] | 63 [32 to 85] | 64 [32 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 23 | 52
  Male | 130 | 146 | 276

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (24-month Rate Reported)
Description: Survival time is defined as time from randomization to date of death from any cause and is estimated by the Kaplan-Meier method. Patients last known to be alive are censored at the date of last contact. This analysis was planned to occur after at least 281 deaths have been observed, unless an early stopping rule was satisfied.
Time Frame: From randomization to last follow-up. Analysis was planned to occur after at least 281 deaths had been observed. Maximum follow-up at time of analysis was 74.5 months.
Population: Eligible patients [We have defined "completed" as patients who have data available for analysis]
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Chemoradiation + Cetuximab | Chemoradiation
Number analyzed (Participants) | 159 | 169
percentage of participants | 44.9 [36.9 to 52.5] | 44.0 [36.4 to 51.4]
Statistical Analysis 1: Comparison: Chemoradiation + Cetuximab vs Chemoradiation; The sample size was based on the primary hypothesis of a 29% reduction in the hazard rate of death with cetuximab, corresponding to an increase in 2-year overall survival (OS) from 41% to 53% and a hazard ratio (λ[exp]/λ[cont]) of 0.71 in favor of the cetuximab arm. Assuming an exponential distribution and constant hazards, 400 patients were required to reach 281 OS events, with 80% statistical power, a 1-sided α of 0.025, 4.5 years of accrual, 2 years of follow-up, and 4 interim analyses; Test type: Superiority; p = 0.47, Log Rank; Hazard Ratio (HR) = 0.90, 95% CI 2-sided [0.70 to 1.16]

2. Secondary Outcome: Local Failure (24-month Rate Reported)
Description: Local failure (LF) was defined as residual cancer on posttreatment biopsy findings or biopsy-proven recurrent primary disease and local failure time was measured from randomization to failure or last follow-up. Nonprotocol surgery to the primary site with gross residual disease was considered a LF as of the surgery date. Patients with no viable disease or microscopic residual disease at nonprotocol surgery were censored for LF as of the surgery date. Local failure was estimated by the cumulative incidence method with death considered a competing risk.
Time Frame: as for outcome 1
Population: All eligible patients
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Chemoradiation + Cetuximab | Chemoradiation
Number analyzed (Participants) | 159 | 169
percentage of participants | 47 [38.3 to 56.6] | 48.8 [40.8 to 57.5]
Statistical Analysis 1: Comparison: Chemoradiation + Cetuximab vs Chemoradiation; Test type: Superiority; p = 0.65, Log Rank; One-sided significance level = 0.025; Hazard Ratio (HR) = 0.92, 95% CI 2-sided [0.66 to 1.28]

3. Secondary Outcome: Percentage of Patients With Acute Grade 4 or 5 Non-hematologic Treatment-related Adverse Events
Description: Adverse events (AE) are graded using CTCAE v3.0. Grade refers to the severity of the AE. The CTCAE v3.0 assigns Grades 1 through 5 with unique clinical descriptions of severity for each AE based on this general guideline: Grade 1 Mild AE, Grade 2 Moderate AE, Grade 3 Severe AE, Grade 4 Life-threatening or disabling AE, Grade 5 Death related to AE
Time Frame: From start of treatment to 90 days from end of treatment
Population: Eligible patients who started study treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Chemoradiation + Cetuximab | Chemoradiation
Number analyzed (Participants) | 153 | 166
percentage of participants | 15.7 [10.8 to 22.3] | 7.8 [4.6 to 12.9]

4. Secondary Outcome: Endoscopic Complete Response Rate
Description: All patients were to undergo a repeat endoscopy (EUS) 6-8 weeks after the completion of chemoradiation. At the time of EUS a visual inspection of the site of the original primary disease would be documented. Those patients found to be free of disease were NOT required to undergo repeat biopsy. These patients would be scored as clinical complete responses (cCR). Patients deemed to have residual disease or suspicion of residual disease would undergo a biopsy in order to pathologically confirm findings. Any patient with pathologically confirmed residual disease would be scored as a local failure. Patients who were pathologically proven to have no evidence of disease would be scored as cCRs.
Time Frame: From randomization to 6-8 weeks after completion of chemoradiation (11-14 weeks)
Population: Eligible patients who started study treatment and had an endoscopy performed
Measure: Number; unit: percentage of participants
Arm/Group | Chemoradiation + Cetuximab | Chemoradiation
Number analyzed (Participants) | 144 | 159
percentage of participants | 56.3 | 57.9
Statistical Analysis 1: Comparison: Chemoradiation + Cetuximab vs Chemoradiation; Test type: Superiority; p = 0.66, Fisher Exact; One-sided significance level = 0.025

5. Secondary Outcome: Percentage of Patients With Improvement in the Functional Assessment of Cancer Therapy - Esophagus (FACT-E) Esophageal Cancer Subscale (ECS) Subscale After Treatment
Description: The ECS is a 17-item self-report instrument designed to measure multidimensional quality of life in patients with esophagus cancer. It is to be administered with the Functional Assessment of Cancer Therapy - General (FACT-G). There are 5 responses options, with 0=Not a lot and 4=Very much. All items are added together to obtain a total score which ranges from 0-68. Certain items must be reversed before it is added by subtracting the response from 4. It requires at least 50% of the items to be completed while the overall response rate of the FACT-E including the FACT-G must be greater than 80%. If items are missing, the subscale scores can be prorated. A higher score indicated better QOL. Improvement in FACT-E score is defined as an increase from baseline score of at least 5 points.
Time Frame: Baseline, 6-8 weeks after completion of chemoradiation , 1 year and 2 years from treatment start.
Population: Patients who consented to collection of patient reported outcomes and quality of life (PRO-QOL) data and had FACT-E scores at baseline and corresponding timepoint
Measure: Number; unit: percentage of participants
Arm/Group | Chemoradiation + Cetuximab | Chemoradiation
Number analyzed (Participants) | 124 | 137
percentage of participants
  6-8 weeks post-treatment: number analyzed (Participants) | 89 | 76
  6-8 weeks post-treatment | 36.8 | 52.8
  1 year: number analyzed (Participants) | 57 | 58
  1 year | 45.6 | 48.3
  2 years: number analyzed (Participants) | 32 | 34
  2 years | 61.3 | 44.1
Statistical Analysis 1: Comparison: Chemoradiation + Cetuximab vs Chemoradiation; 6-8 weeks post-treatment; Test type: Superiority; p = 0.04, Chi-squared; Two-sided significance level = 0.05
Statistical Analysis 2: Comparison: Chemoradiation + Cetuximab vs Chemoradiation; 1 year; Test type: Superiority; p = 0.77, Chi-squared; Two-sided significance level = 0.05
Statistical Analysis 3: Comparison: Chemoradiation + Cetuximab vs Chemoradiation; 2 years; Test type: Superiority; p = 0.17, Chi-squared; Two-sided significance level = 0.05

6. Secondary Outcome: Quality-adjusted Survival (Using EQ-5D), Only if Primary Hypothesis is Supported
Time Frame: Baseline, 6-8 weeks after completion of chemoradiation, 1 year and 2 years from treatment start.
Population: The protocol states that this study endpoint will be addressed ONLY if primary outcome results are positive, i.e. support the primary hypothesis of this study. The primary hypothesis was not supported therefore no patients were analyzed for this outcome measure.
Arm/Group | Chemoradiation + Cetuximab | Chemoradiation
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: All patients who started study treatment are included, including ineligible patients. (Therefore this patient group differs from Outcome Measure 3, which is restricted to eligible patients.) Subjects experiencing more than one of a given adverse event are counted only once for that adverse event.
Groups:
- Chemoradiation + Cetuximab: External beam radiation therapy (RT) with concurrent weekly paclitaxel, and cisplatin, a
Arm/Group | Chemoradiation + Cetuximab | Chemoradiation
Serious Adverse Events (participants affected / at risk) | 88/162 | 88/173
Other Adverse Events (participants affected / at risk) | 156/162 | 169/173
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Chemoradiation + Cetuximab (N=162) | Chemoradiation (N=173)
Blood disorder (Blood and lymphatic system disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 4 | 3
Hemoglobin decreased (Blood and lymphatic system disorders) | 10 | 10
Hemolysis (Blood and lymphatic system disorders) | 0 | 1
Arrhythmia (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 7 | 0
Atrial flutter (Cardiac disorders) | 1 | 2
Cardiac disorder (Cardiac disorders) | 3 | 1
Cardiac pain (Cardiac disorders) | 1 | 0
Left ventricular failure (Cardiac disorders) | 0 | 1
Myocardial ischemia (Cardiac disorders) | 3 | 2
Pericardial effusion (Cardiac disorders) | 2 | 0
Pericarditis (Cardiac disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 2
Supraventricular tachycardia (Cardiac disorders) | 0 | 1
Ventricular arrhythmia (Cardiac disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 4 | 4
Acquired tracheo-oesophageal fistula (Gastrointestinal disorders) | 1 | 3
Colitis (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 1
Diarrhea (Gastrointestinal disorders) | 10 | 6
Duodenal obstruction (Gastrointestinal disorders) | 0 | 1
Duodenal perforation (Gastrointestinal disorders) | 1 | 0
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 1
Dysphagia (Gastrointestinal disorders) | 13 | 13
Enteritis (Gastrointestinal disorders) | 1 | 0
Esophageal hemorrhage (Gastrointestinal disorders) | 2 | 3
Esophageal mucositis (Gastrointestinal disorders) | 0 | 2
Esophageal pain (Gastrointestinal disorders) | 5 | 8
Esophageal perforation (Gastrointestinal disorders) | 1 | 1
Esophageal stenosis (Gastrointestinal disorders) | 0 | 2
Esophageal ulcer (Gastrointestinal disorders) | 1 | 1
Esophageal varices hemorrhage (Gastrointestinal disorders) | 0 | 1
Esophagitis (Gastrointestinal disorders) | 13 | 12
Gastric hemorrhage (Gastrointestinal disorders) | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 2
Gastro-intestinal fistula (Gastrointestinal disorders) | 0 | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 2 | 0
Jejunal perforation (Gastrointestinal disorders) | 0 | 1
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 1
Malabsorption (Gastrointestinal disorders) | 1 | 0
Mucositis oral (Gastrointestinal disorders) | 3 | 1
Nausea (Gastrointestinal disorders) | 17 | 14
Obstruction gastric (Gastrointestinal disorders) | 0 | 2
Oral pain (Gastrointestinal disorders) | 0 | 1
Rectal hemorrhage (Gastrointestinal disorders) | 1 | 0
Stomach pain (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 3
Vomiting (Gastrointestinal disorders) | 16 | 12
Chest pain (General disorders) | 3 | 3
Chills (General disorders) | 1 | 0
Death (General disorders) | 4 | 1
Disease progression (General disorders) | 1 | 0
Fatigue (General disorders) | 13 | 8
Fever (General disorders) | 5 | 5
General symptom (General disorders) | 2 | 0
Pain (General disorders) | 2 | 1
Sudden death (General disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Hepatic hemorrhage (Hepatobiliary disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 5 | 2
Immune system disorder (Immune system disorders) | 1 | 0
Abdominal infection (Infections and infestations) | 1 | 0
Appendicitis perforated (Infections and infestations) | 1 | 0
Bladder infection (Infections and infestations) | 1 | 1
Catheter related infection (Infections and infestations) | 0 | 1
Gallbladder infection (Infections and infestations) | 0 | 1
Gastric infection (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 2 | 2
Jejunal infection (Infections and infestations) | 1 | 0
Joint infection (Infections and infestations) | 1 | 0
Mucosal infection (Infections and infestations) | 1 | 0
Opportunistic infection (Infections and infestations) | 1 | 0
Peritoneal infection (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 6 | 3
Sepsis (Infections and infestations) | 2 | 3
Skin infection (Infections and infestations) | 1 | 0
Stoma site infection (Infections and infestations) | 1 | 0
Wound infection (Infections and infestations) | 1 | 1
Anastomotic leak (Injury, poisoning and procedural complications) | 0 | 1
Esophageal anastomotic leak (Injury, poisoning and procedural complications) | 0 | 1
Prolonged intubation after pulmonary resection (>24 hrs after surgery) (Injury, poisoning and procedural complications) | 0 | 1
Radiation recall reaction (dermatologic) (Injury, poisoning and procedural complications) | 2 | 0
Vascular access complication (Injury, poisoning and procedural complications) | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1
Activated partial thromboplastin time prolonged (Investigations) | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1
Alkaline phosphatase increased (Investigations) | 1 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 1
Cardiac troponin I increased (Investigations) | 0 | 1
Hyperbilirubinemia (Investigations) | 0 | 1
INR increased (Investigations) | 0 | 1
Leukopenia (Investigations) | 13 | 11
Lymphopenia (Investigations) | 3 | 4
Neutrophil count decreased (Investigations) | 13 | 7
Platelet count decreased (Investigations) | 4 | 5
Weight loss (Investigations) | 7 | 9
Anorexia (Metabolism and nutrition disorders) | 6 | 4
Dehydration (Metabolism and nutrition disorders) | 32 | 24
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 2
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 0
Hypernatremia (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 4 | 3
Hypocalcemia (Metabolism and nutrition disorders) | 5 | 2
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 3 | 3
Hypomagnesemia (Metabolism and nutrition disorders) | 6 | 5
Hyponatremia (Metabolism and nutrition disorders) | 5 | 3
Hypophosphatemia (Metabolism and nutrition disorders) | 4 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Muscle weakness (Musculoskeletal and connective tissue disorders) | 3 | 1
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 4
Extrapyramidal disorder (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Ischemia cerebrovascular (Nervous system disorders) | 2 | 0
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 2 | 7
Confusion (Psychiatric disorders) | 2 | 5
Renal failure (Renal and urinary disorders) | 1 | 0
Urogenital disorder (Renal and urinary disorders) | 0 | 1
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Hiccough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Acne (Skin and subcutaneous tissue disorders) | 4 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0
Rash desquamating (Skin and subcutaneous tissue disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 3
Hypotension (Vascular disorders) | 5 | 4
Peripheral ischemia (Vascular disorders) | 1 | 0
Thrombosis (Vascular disorders) | 5 | 7
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Chemoradiation + Cetuximab (N=162) | Chemoradiation (N=173)
Hemoglobin decreased (Blood and lymphatic system disorders) | 88 | 87
Pericardial effusion (Cardiac disorders) | 8 | 2
Abdominal pain (Gastrointestinal disorders) | 21 | 20
Constipation (Gastrointestinal disorders) | 57 | 47
Diarrhea (Gastrointestinal disorders) | 54 | 35
Dry mouth (Gastrointestinal disorders) | 9 | 9
Dyspepsia (Gastrointestinal disorders) | 25 | 20
Dysphagia (Gastrointestinal disorders) | 79 | 89
Esophageal pain (Gastrointestinal disorders) | 20 | 24
Esophageal stenosis (Gastrointestinal disorders) | 7 | 12
Esophagitis (Gastrointestinal disorders) | 47 | 49
Gastrointestinal disorder (Gastrointestinal disorders) | 10 | 5
Mucositis oral (Gastrointestinal disorders) | 28 | 9
Nausea (Gastrointestinal disorders) | 87 | 96
Vomiting (Gastrointestinal disorders) | 47 | 60
Chest pain (General disorders) | 12 | 15
Edema limbs (General disorders) | 13 | 11
Fatigue (General disorders) | 108 | 108
Fever (General disorders) | 17 | 17
Pain (General disorders) | 10 | 16
Hypersensitivity (Immune system disorders) | 8 | 6
Dermatitis radiation (Injury, poisoning and procedural complications) | 31 | 43
Radiation recall reaction (dermatologic) (Injury, poisoning and procedural complications) | 23 | 7
Alanine aminotransferase increased (Investigations) | 15 | 11
Alkaline phosphatase increased (Investigations) | 12 | 16
Aspartate aminotransferase increased (Investigations) | 23 | 18
Creatinine increased (Investigations) | 24 | 26
Hyperbilirubinemia (Investigations) | 5 | 9
Laboratory test abnormal (Investigations) | 8 | 10
Leukopenia (Investigations) | 98 | 84
Lymphopenia (Investigations) | 29 | 31
Neutrophil count decreased (Investigations) | 59 | 53
Platelet count decreased (Investigations) | 60 | 63
Weight loss (Investigations) | 107 | 97
Anorexia (Metabolism and nutrition disorders) | 57 | 39
Dehydration (Metabolism and nutrition disorders) | 47 | 37
Hyperglycemia (Metabolism and nutrition disorders) | 53 | 54
Hyperkalemia (Metabolism and nutrition disorders) | 5 | 10
Hypoalbuminemia (Metabolism and nutrition disorders) | 55 | 50
Hypocalcemia (Metabolism and nutrition disorders) | 52 | 35
Hypokalemia (Metabolism and nutrition disorders) | 45 | 30
Hypomagnesemia (Metabolism and nutrition disorders) | 75 | 51
Hyponatremia (Metabolism and nutrition disorders) | 49 | 53
Back pain (Musculoskeletal and connective tissue disorders) | 12 | 16
Muscle weakness (Musculoskeletal and connective tissue disorders) | 14 | 11
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 | 8
Dizziness (Nervous system disorders) | 20 | 24
Headache (Nervous system disorders) | 16 | 15
Peripheral sensory neuropathy (Nervous system disorders) | 20 | 19
Taste alteration (Nervous system disorders) | 25 | 20
Anxiety (Psychiatric disorders) | 9 | 14
Depression (Psychiatric disorders) | 15 | 11
Insomnia (Psychiatric disorders) | 18 | 18
Cough (Respiratory, thoracic and mediastinal disorders) | 36 | 33
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 28 | 37
Hiccough (Respiratory, thoracic and mediastinal disorders) | 6 | 9
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 15 | 10
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 10 | 6
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 | 9
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 13 | 9
Acne (Skin and subcutaneous tissue disorders) | 93 | 4
Alopecia (Skin and subcutaneous tissue disorders) | 27 | 12
Dry skin (Skin and subcutaneous tissue disorders) | 40 | 9
Pruritus (Skin and subcutaneous tissue disorders) | 30 | 11
Rash desquamating (Skin and subcutaneous tissue disorders) | 33 | 15
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 8 | 6
Hypotension (Vascular disorders) | 20 | 18

LIMITATIONS AND CAVEATS:
After a United Kingdom trial failed to show a benefit for cetuximab, accrual was suspended and the 3rd planned interim analysis done. After discussions with the Data Monitoring Committee, the study permanently closed to accrual on 2/8/2013.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI's are required to abide by the sponsor's publication guidelines which require review by coauthors and subsequent review and approval by the sponsor.